CLINICAL TRIAL: NCT05925504
Title: Safety and Efficacy Study of the Tapering Dose of Luspatercept in Patients With Lower-risk Myelodysplastic Syndromes
Brief Title: The Tapering Dose of Luspatercept in Patients With Lower-risk Myelodysplastic Syndromes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Beijing Health Alliance Charitable Foundation (Unknown)
Responsible Party: Principal Investigator, Gao Zhen, Physician of Regenerative Medical Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lusp-MDS
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Lower Risk MDS Per IPSS-R
MeSH Terms: interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luspatercept (Experimental): open-label, single-arm
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — The starting dose is 1.75mg/kg once every 3 weeks by subcutaneous injection. For rapid hemoglobin rise after 2 consecutive doses at the 1.75mg/kg starting dose, decrease the dose of Luspatercept or interrupt treatment. Otherwise, continue treatment with the dose of 1.75mg/kg once every 3 weeks.

SUMMARY:
This is a prospective, single center, single-arm, phase 2 study. The aim of this study is to evaluate the efficacy and safety of Luspatercept for Patients with Lower-risk Myelodysplastic Syndromes (MDS).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years
* Subject has diagnosis of MDS according to WHO classification that meets IPSS-R score ≤3.5
* Hemoglobin < 100g/L at baseline
* Refractory or intolerant to prior ESA treatment or EPO≥500U/L
* ECOG performance status ≤2
* Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

* Platelet counts < 50 x 10^9/L
* Previously treated with either luspatercept or sotatercept
* Use any of the following prior to this study

  * Immunomodulatory drugs such as lenalidomide [IMiD] for ≥4 weeks
  * Immunosuppressive therapy [IST] for ≥4 weeks
  * Demethylating agents [HMA] ≥ 1 cycle of treatment
* MDS associated with del 5q cytogenetic abnormality
* Secondary MDS, i.e. MDS that is known to have arisen as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases.
* Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding.
* Prior allogeneic or autologous stem cell transplant.
* Prior history of malignancies, other than MDS, unless the subject is free of the disease (including completion of any active or adjuvant treatment for prior malignancy) for ≥ 5 years. However, subjects with the following history/concurrent conditions are allowed: basal or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasia, carcinoma in situ of the cervix or other indolent tumors.
* Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment), known human immunodeficiency virus (HIV), known evidence of active infectious hepatitis B, and/or known evidence of active hepatitis C.
* Clinically significant cardiac disease, including any of the follow: uncontrolled angina pectoris, myocardial infarction, unstable cardiac arrhythmias, congestive heart failure and New York Heart Association (NYHA) grade 2-4 cardiac failure.
* Abnormal liver function: two consecutive examinations with an interval of ≥1 week suggest that ALT and AST are 2.5 times higher than the upper limit of normal values
* Renal impairment: creatinine clearance <60ml/min
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study, including clinically significant cardiac diseases, refractory hypertension, metabolic disorders and other diseases that seriously affect the function of the gastrointestinal tract.
* Had a history of any psychiatric diseases, cerebrovascular disease or cognitive sequelae of head injury.
* Major surgery within 8 weeks prior to this study. Subjects must be completely recovered from any previous surgery prior to this study.
* Received attenuated vaccine in 4 weeks before enrollment.
* Participation in another clinical trial within 4 weeks before the start of this trial.
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the luspatercept.
* Pregnant or breast-feeding patients
* Patients considered to be ineligible for the study by the investigator for reasons other than the above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving hematologic improvement - erythroids (HI-E) according to IWG 2006 criteria | within 12 weeks

SECONDARY OUTCOMES:
Proportion of subjects achieving RBC-TI according to IWG 2006 criteria | within 12 weeks
Median time to HI-E or RBC-TI | within 12 weeks
Mean change in serum ferritin | within 12 weeks
Incidence of the adverse event | within 12 weeks
  Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Medicine Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No